CLINICAL TRIAL: NCT01004978
Title: A Phase III Randomized, Double-Blind Trial of Chemoembolization With or Without Sorafenib in Unresectable Hepatocellular Carcinoma (HCC) in Patients With and Without Vascular Invasion
Brief Title: Chemoembolization With or Without Sorafenib Tosylate in Treating Patients With Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-01981; NCI-2011-01981 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E1208; 10-00544; CDR0000657952; E1208 (Other: ECOG-ACRIN Cancer Research Group); E1208 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH)
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2023-02-17 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma; Unresectable Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Doxorubicin; Magnetic Resonance Spectroscopy; Mitomycin; Mitozytrex; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (sorafenib tosylate and TACE) (Experimental): Patients receive sorafenib tosylate PO BID in the absence of disease progression or unacceptable toxicity. Beginning within 2 weeks after a stable dose of sorafenib tosylate is reached, patients undergo TACE comprising doxorubicin hydrochloride, mitomycin C, and cisplatin (closed to accrual as of 10/1/2010); conventional chemoembolization comprising doxorubicin hydrochloride only; or chemoembolization comprising doxorubicin-eluting beads. Treatment with TACE repeats approximately every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and MRI on study.
  Interventions: Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Drug: Doxorubicin-Eluting Beads; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Other: Pharmacological Study; Drug: Sorafenib Tosylate
- Arm II (placebo and TACE) (Active Comparator): Patients receive placebo PO BID in the absence of disease progression or unacceptable toxicity. Beginning within 2 weeks after a stable dose of placebo is reached, patients undergo TACE as in Arm I. Patients also undergo CT and MRI on study.
  Interventions: Drug: Cisplatin; Procedure: Computed Tomography; Drug: Doxorubicin Hydrochloride; Drug: Doxorubicin-Eluting Beads; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Other: Pharmacological Study; Other: Placebo Administration

INTERVENTIONS:
Drug: Cisplatin — Undergo TACE
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Doxorubicin Hydrochloride — Undergo TACE
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Doxorubicin-Eluting Beads — Undergo TACE
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mitomycin — Undergo TACE
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
Other: Pharmacological Study — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II (placebo and TACE)
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
  Arms: Arm I (sorafenib tosylate and TACE)

SUMMARY:
This randomized phase III trial studies chemoembolization and sorafenib tosylate to see how well they work compared with chemoembolization alone in treating patients with liver cancer that cannot be removed by surgery. Drugs used in chemotherapy, such as doxorubicin hydrochloride, mitomycin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Chemoembolization kills tumor cells by carrying drugs directly into blood vessels near the tumor and then blocking the blood flow to allow a higher concentration of the drug to reach the tumor for a longer period of time. Kinase inhibitors, such as sorafenib tosylate may stop the growth of tumor cells by blocking the action of an abnormal protein that signals cancer cells to multiply. It is not yet known whether giving chemoembolization together with sorafenib tosylate is more effective than chemoembolization alone in treating patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival (PFS) of chemoembolization alone to sorafenib (sorafenib tosylate) in combination with chemoembolization.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) of chemoembolization alone to sorafenib in combination with chemoembolization.

II. To evaluate extra-hepatic versus intra-hepatic patterns of failure. III. To determine the rates of toxicity related to sorafenib in combination with chemoembolization.

TERTIARY OBJECTIVES:

I. To analyze the pharmacogenetic and pharmacokinetic properties of sorafenib including angiogenesis, monooxygenases, polymorphisms and multidrug resistance (MDR).

II. Eastern Cooperative Oncology Group (ECOG)-American College of Radiology Imaging Network (ACRIN) secondary imaging objective: site versus (vs.) central evaluation of PFS.

III. To determine the inter-reader concordance for response characterization at four and eight months by the European Association for the Study of Liver (EASL) criteria.

IV. To determine the value of objective tumor response at four and eight months by the EASL criteria to predict PFS (by Response Evaluation Criteria in Solid Tumors [RECIST]) and OS.

V. To evaluate the effects of intra-hepatic vs. extra-hepatic progression on OS.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive sorafenib tosylate orally (PO) twice daily (BID) in the absence of disease progression or unacceptable toxicity. Beginning within 2 weeks after a stable dose of sorafenib tosylate is reached, patients undergo transarterial chemoembolization (TACE) comprising doxorubicin hydrochloride, mitomycin C, and cisplatin (closed to accrual as of 10/1/2010); conventional chemoembolization comprising doxorubicin hydrochloride only; or chemoembolization comprising doxorubicin-eluting beads. Treatment with TACE repeats approximately every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and magnetic resonance imaging (MRI) on study.

ARM II: Patients receive placebo PO BID in the absence of disease progression or unacceptable toxicity. Beginning within 2 weeks after a stable dose of placebo is reached, patients undergo TACE as in Arm I. Patients also undergo CT and MRI on study.

MAINTENANCE THERAPY: After completion of chemoembolization, patients receive sorafenib tosylate or placebo as in Arm I and II in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of hepatocellular carcinoma by at least one criterion listed below:

  * Histologically confirmed
  * Magnetic resonance imaging (MRI) or computerized tomography (CT) consistent with liver cirrhosis AND at least one solid liver lesion > 2 cm with early enhancement and delayed enhancement washout regardless of alpha-feto protein levels (AFP)
  * AFP > 400 ng/mL AND evidence of at least one solid liver lesion > 2 cm regardless of specific imaging characteristics on CT or MRI
* Patients must have hepatocellular carcinoma (HCC) limited to the liver; there must be no clinical or radiographic evidence of extrahepatic HCC
* Portal lymphadenopathy IS permitted for patients with hepatitis B virus (HBV) or hepatitis C virus (HCV) - as lymphadenopathy is commonly associated with hepatitis unrelated to malignancy
* Staging CT of the chest and CT or MRI of the abdomen and pelvis must have been completed within 4 weeks of study registration
* Patients must have measurable disease constituting < 50% of liver parenchyma within 4 weeks of registration
* Patients may not have ascites detectable on physical examination
* Patients must not be candidates for curative resection, orthotopic liver transplantation, or radiofrequency ablation (RFA)
* Patients may have been treated with RFA in the past, but no sooner than 4 weeks before study registration
* Patients may have undergone previously attempted curative liver resection
* Patients may NOT have been previously treated with brachytherapy such as yttrium-90 microsphere
* Patients may NOT have been previously treated with sorafenib, chemoembolization, or systemic chemotherapy including cytotoxic agents or molecularly targeted agents
* Branch portal vein invasion by tumor is permitted but patients with main portal vein invasion by tumor are not eligible
* Patients must have Child-Pugh score of A or B7 within 4 weeks prior to study registration
* Serum total bilirubin =< 2.0 mg/dL
* Alkaline phosphatase < 5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 5 x ULN
* Serum creatinine =< 1.5 mg/dL
* Platelet count >= 50,000/mm^3
* Patients must not have any evidence of bleeding diathesis or active gastrointestinal bleeding
* Patients must have no clinical signs of heart failure and meet New York Heart Association functional classification I or II defined as:

  * Class I - patients with no limitation of activities; they suffer no symptoms from ordinary activities
  * Class II - patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have a life expectancy of at least 3 months
* Patients must not be known to be human immunodeficiency virus (HIV) positive
* Patients must not have other uncontrolled intercurrent illnesses excluding HBV or HCV, including, but not limited to: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/addictive disorders that would limit compliance with study requirements

  * Uncontrolled hypertension is defined as optimally treated baseline blood pressure that exceeds 150/90 mm Hg
* Patients must not be taking cytochrome P450 enzyme inducing drugs
* Age >= 18 years
* Women must not be pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception
* Patients must not have an allergy to iodine or gadolinium contrast that cannot be safely controlled with premedication
* Patient must be able to swallow pills, as study medications cannot be crushed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2009-10-28 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al B Benson, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (281):
- United States (281):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Marin Cancer Care Inc, Greenbrae, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Veterans Affairs Medical Center -Washington DC, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMITA Health Adventist Medical Center, La Grange, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Administration, Columbia, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Veteran Affairs New York Harbor Healthcare System-Brooklyn Campus, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Mount Sinai Union Square, New York, New York
  - Veterans Affairs New York Harbor Healthcare System-Manhattan Campus, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study activated on October 28, 2009 and closed to accrual on November 19, 2014 due to poor enrollment. A total of 235 patients were randomized.
Groups:
- Arm A (Sorafenib and TACE): Patients receive sorafenib tosylate at 400mg PO BID in the absence of disease progression or unacceptable toxicity. Beginning within 2 weeks after a stable dose of sorafenib tosylate is reached, patients undergo TACE comprising doxorubicin hydrochloride, mitomycin C, and cisplatin (this option may only be utilized for patients registered prior to addendum #3); conventional chemoembolization comprising doxorubicin hydrochloride only; or chemoembolization comprising LC bead and doxorubicin. Treatment with TACE repeats approximately every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (Placebo and TACE): Patients receive placebo PO BID in the absence of disease progression or unacceptable toxicity. Beginning within 2 weeks after a stable dose of placebo is reached, patients undergo TACE as in Arm A.
Period: Overall Study
Arm/Group | Arm A (Sorafenib and TACE) | Arm B (Placebo and TACE)
Started | 118 | 117
Completed | 0 (Treatment was given until disease progression.) | 0 (Treatment was given until disease progression.)
Not Completed | 118 | 117
Not completed — Disease progression | 31 | 48
Not completed — Adverse Event | 42 | 22
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 16 | 16
Not completed — Alternative therapy | 4 | 8
Not completed — Physician Decision | 6 | 3
Not completed — Other complicating disease | 2 | 2
Not completed — Protocol Violation | 2 | 3
Not completed — Non-compliance | 3 | 2
Not completed — Ineligible | 1 | 0
Not completed — Unblinded | 0 | 1
Not completed — Performance status worsening | 0 | 1
Not completed — Never started treatment | 8 | 9

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Sorafenib and TACE) | Arm B (Placebo and TACE) | Total
Number analyzed (Participants) | 118 | 117 | 235
Age, Continuous [Median (Full Range); unit: years] | 62.1 [41 to 82] | 64.1 [32 to 88] | 62.8 [32 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 104 | 101 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 14 | 30
  Not Hispanic or Latino | 99 | 98 | 197
  Unknown or Not Reported | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 14 | 13 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 22 | 51
  White | 71 | 78 | 149
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined to be the time from randomization to progression or death without evidence of progression. For cases without documentation of progression, follow-up will be censored at the date of last disease assessment without progression, unless death occurs within 4 months following the date last known progression-free, in which case the death will be counted as an event.
  Progression is assessed per Solid Tumor Response Criteria (RECIST) and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions.
Time Frame: Assessed 4 months after first chemoembolization, 8 months after first chemoembolization, then every 8 weeks, up to 4 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Sorafenib and TACE) | Arm B (Placebo and TACE)
Number analyzed (Participants) | 118 | 117
months | 9.3 [6.8 to 11.9] | 8.4 [5.4 to 10.9]
Statistical Analysis 1: Comparison: Arm A (Sorafenib and TACE) vs Arm B (Placebo and TACE); Test type: Superiority; p = 0.4, Cochran-Mantel-Haenszel — one-sided p-value

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as time from randomization to death from any cause, censoring cases who had not died at the date last known alive.
Time Frame: Assessed every 3 months for 2 years and then every 6 months for 2 years
Population: All randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Sorafenib and TACE) | Arm B (Placebo and TACE)
Number analyzed (Participants) | 118 | 117
months | 19.8 [16.8 to 23.7] | 19.9 [13.5 to 27.2]
Statistical Analysis 1: Comparison: Arm A (Sorafenib and TACE) vs Arm B (Placebo and TACE); Test type: Superiority; p = 0.76, Log Rank

3. Secondary Outcome: Progression-free Survival (PFS) Among Patients With Extra-hepatic Progression
Description: PFS is defined to be the time from randomization to progression or death without evidence of progression.
  Progression is assessed per Solid Tumor Response Criteria (RECIST) and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions.
  For patients with progressive disease, the progression was classified as either intra- or extra-hepatic or both intra- and extra-hepatic. Patients with both intra- and extra-hepatic progression were considered as having extra-hepatic progression. This analysis was performed among patients with extra-hepatic progression.
Time Frame: as for outcome 1
Population: Only patients with extra-hepatic progression (as well as those with both intra- and extra-hepatic progression) are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Sorafenib and TACE) | Arm B (Placebo and TACE)
Number analyzed (Participants) | 19 | 11
months | 6.83 [3.7 to 15.7] | 5.6 [5.0 to 9.7]

4. Secondary Outcome: Progression-free Survival (PFS) Among Patients With Intra-hepatic Progression
Description: PFS is defined to be the time from randomization to progression or death without evidence of progression.
  Progression is assessed per Solid Tumor Response Criteria (RECIST) and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions.
  For patients with progressive disease, the progression was classified as either intra- or extra-hepatic or both intra- and extra-hepatic. This analysis was performed among patients with intra-hepatic progression.
Time Frame: as for outcome 1
Population: Only patients with intra-hepatic progression are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Sorafenib and TACE) | Arm B (Placebo and TACE)
Number analyzed (Participants) | 53 | 64
months | 8.5 [5.8 to 11.1] | 7.8 [4.9 to 10.7]

5. Other Pre Specified Outcome: Pharmacogenetic and Pharmacokinetic Properties of Sorafenib Including Angiogenesis, Monooxygenases, Polymorphisms and Multidrug Resistance Mutation (MDR)
Description: This analysis will be performed across a few ECOG-ACRIN studies of sorafenib to evaluate the association between genotypes that are related with sorafenib activity and clinical outcomes.
Time Frame: Assessed at baseline, days 1, 8 and 15 of cycle 1 sorafenib, 3-5 days prior to 2nd and 3rd TACE
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Inter-reader Concordance for Response by EASL (European Association for the Study of the Liver) Criteria
Description: Response was determined using the European Association for the Study of the Liver (EASL) criteria, which was recommended as an alternative to RECIST for grading therapeutic response of advanced hepatocellular carcinoma (HCC). The EASL criteria use the longest dimension of enhancing tumor as the primary metric for gauging tumor response. The Kappa statistics will be applied to assess agreement between readers.
Time Frame: at 4 months and 8 months Assessed at 4 months and 8 months following initial chemoembolization
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Association Between Objective Tumor Response by EASL Criteria and PFS as Well as OS
Description: PFS is defined to be the time from randomization to progression or death without evidence of progression. For cases without documentation of progression, follow-up will be censored at the date of last disease assessment without progression, unless death occurs within 4 months following the date last known progression-free, in which case the death will be counted as an event.
  Progression is assessed per Solid Tumor Response Criteria (RECIST) and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions.
  OS is defined as time from randomization to death or date last known alive. Response is assessed at 4 and 8 months by EASL criteria.
Time Frame: as for outcome 1
Reporting Status: Not Posted

8. Other Pre Specified Outcome: To Evaluate the Effects of Intra-hepatic vs. Extra-hepatic Progression on OS.
Description: Progression is assessed per Solid Tumor Response Criteria (RECIST) and defined as at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s), and/or unequivocal progression of existing nontarget lesions.
  For patients with progressive disease, the progression was classified as either intra- or extra-hepatic or both intra- and extra-hepatic.
  OS is defined as the time from randomization to death or date last known alive.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, and then every 6 months up to 4 years
Description: Adverse events were assessed among all treated patients. All-cause mortality was evaluated among all randomized patients.
Groups:
- Arm A (Sorafenib and TACE): Patients receive sorafenib tosylate PO BID in the absence of disease progression or unacceptable toxicity. Beginning within 2 weeks after a stable dose of sorafenib tosylate is reached, patients undergo TACE comprising doxorubicin hydrochloride, mitomycin C, and cisplatin (this option may only be utilized for patients registered prior to addendum #3); conventional chemoembolization comprising doxorubicin hydrochloride only; or chemoembolization comprising LC bead and doxorubicin. Treatment with TACE repeats approximately every 4 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Sorafenib and TACE) | Arm B (Placebo and TACE)
All-Cause Mortality (participants affected / at risk) | 85/118 | 88/117
Serious Adverse Events (participants affected / at risk) | 65/110 | 41/108
Other Adverse Events (participants affected / at risk) | 22/110 | 21/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sorafenib and TACE) (N=110) | Arm B (Placebo and TACE) (N=108)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 5 | 3
Gait disturbance (General disorders) | 2 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 11 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 7
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 2
Esophageal hemorrhage (Gastrointestinal disorders) | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic hemorrhage (Hepatobiliary disorders) | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Peripheral nerve infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 7 | 8
Alkaline phosphatase increased (Investigations) | 2 | 4
Aspartate aminotransferase increased (Investigations) | 15 | 12
Blood bilirubin increased (Investigations) | 9 | 4
Creatinine increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 5 | 0
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Hypertension (Vascular disorders) | 9 | 3
Hypotension (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sorafenib and TACE) (N=110) | Arm B (Placebo and TACE) (N=108)
Anemia (Blood and lymphatic system disorders) | 6 | 11
Fatigue (General disorders) | 15 | 13
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 8 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Diarrhea (Gastrointestinal disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 8 | 8
Platelet count decreased (Investigations) | 9 | 9
Weight loss (Investigations) | 7 | 1
White blood cell decreased (Investigations) | 6 | 2
Anorexia (Metabolism and nutrition disorders) | 9 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT01004978/Prot_SAP_000.pdf